CLINICAL TRIAL: NCT04458935
Title: Retrospective Case Series of Trans-scleral Cryotherapy for Retinal Hemangioblastoma
Status: Active, not recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999920129; 20-EI-N129
Record Dates: First submitted 2020-07-03; First posted 2020-07-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Retinal Hemangioblastoma; Von Hippel-Lindau Disease
Keywords: Vascular Tumor; Vision Loss; Natural History
MeSH Terms: conditions — von Hippel-Lindau Disease; Vascular Neoplasms; Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Participants with retinal hemangioblastoma (RH) managed with trans-scleral cryotherapy at the NIH.

SUMMARY:
Background:

Retinal hemangioblastoma (RH) is a tumor. It grows from the retina in the eye. It can threaten a person s vision. Trans-scleral cryotherapy is used to destroy the tumors and minimize the long-term risks of vision loss. RH is a rare condition, often occurring in people with von Hippel-Lindau disease. There are no clinical trials to study how well the treatment works. Researchers want to study the medical records of people with RH who were treated at the NIH eye clinic to learn more.

Objective:

To analyze clinical data collected over a 20-year span to study consecutive cases of RH managed with trans-scleral cryotherapy at the NIH.

Eligibility:

People who took part in NIH natural history protocols for which cryotherapy of RH was performed as a standard care measure.

Design:

Researchers will collect and study data from participants medical charts. Participants will not be contacted because no new data is needed. Researchers were granted a waiver of informed consent for use of these medical records. To protect patient privacy, participants will be assigned an ID number. Their data will be entered into a spreadsheet in a coded fashion. The key to this code will be kept in a secure file. No patient identifying information will be used in the analysis or the publication....

DETAILED DESCRIPTION:
Study Description: This study is a retrospective review of medical records in the NIH eye clinic. To our knowledge, there has been no report in the current era dedicated to a description of trans-scleral cryotherapy for retinal hemangioblastomas despite its routine use in this setting. This study aims to explore features and outcomes of these cases to better inform best practices.

Objectives: The objective of this study is to perform a retrospective analysis of consecutive cases of retinal hemangioblastoma managed with trans-scleral cryotherapy at the NIH (single center retrospective case series).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participants were enrolled in NEI and non-NEI natural history protocols, but in all cases, cryotherapy was administered as a standard care measure (not as an investigative treatment).
  2. Patients were identified by searching the NIH eye clinic EMR for all of those manifesting one or more retinal hemangioblastomas (with or without associated von Hippel-Lindau disease) treated with cryotherapy.

EXCLUSION CRITERIA:

None

Ages: 7 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data (medical history and images) was collected under NEI and non-NEI natural history protocols allowing administration of standard care measures to participants.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To perform a retrospective analysis of consecutive cases of retinal hemangioblastoma (RH) managed with trans-scleral cryotherapy at the NIH | ongoing
  Some key measures of interest will include treatment outcomes (rate of control of tumors; visual function measures; post-treatment lesion characteristics; sequelae and complications) and association of outcomes with eye and lesion characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No